CLINICAL TRIAL: NCT04270500
Title: The Impact of Physical Exercise on Sleep Quality and Duration in Colorectal Cancer Patients During Prehabilitation Period: A Pilot Study
Brief Title: The Impact of Physical Exercise on Sleep in Colorectal Cancer Patients During Prehabilitation Period
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Montreal General Hospital (Other)
Responsible Party: Principal Investigator, Sender Liberman MD, Principal Investigator, Montreal General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PA-Sleep
Record Dates: First submitted 2020-02-07; First posted 2020-02-17 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Colo-rectal Cancer; Surgery
Keywords: Colo-rectal Cancer; Colo-rectal Surgery; Prehabilitation; Sleep quality; Sleep duration; Physical exercise
MeSH Terms: conditions — Colonic Neoplasms; Sleep Initiation and Maintenance Disorders; Motor Activity

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled pilot trial of patients with colorectal cancer scheduled for major abdominal surgery. The prehabilitation intervention group will be compared with the usual care for an average of 4 weeks before planned surgery. All participants will wear an actigraphy to objectively assess their daily physical activity and their sleep behavior.
  The intervention will last for 4 weeks pre- and 8 weeks post-surgery, for a total of 12 weeks. Site visits will occur weekly before surgery and every 4 weeks after surgery. In that period, weekly phone calls will reinforce compliance and provide tips to help patients adhere to the treatment protocol. A dedicated and specially trained research team lead by a physician, a kinesiologist, a nutritionist and a psychologist will perform the measurements and collect the demographic and surgical details of all the patients, recording daily detailed information of clinical outcomes up to 8 weeks after surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prehabilitation program (Active Comparator): The preoperative period (prehabilitation) represents a more appropriate time than the postoperative period to implement an intervention. Prehabilitation is a process of enhancing an individual's functional capacity before the scheduled surgery, aimed at improving the patient's tolerance to upcoming physiologic stress, by three principal elements: exercise training, nutritional intervention, and psychological support.
  Interventions: Behavioral: Prehabilitation program
- Standard of care (SOC) (No Intervention): Common to both groups as part of the enhanced recovery after surgery (ERAS) protocol as the standard of care in our institution.

INTERVENTIONS:
Behavioral: Prehabilitation program — The preoperative period (prehabilitation) represents a more appropriate time than the postoperative period to implement an intervention. Prehabilitation is a process of enhancing an individual's functional capacity before the scheduled surgery, aimed at improving the patient's tolerance to upcoming physiologic stress, by three principal elements: exercise training, nutritional intervention, and psychological support.
  Arms: Prehabilitation program

SUMMARY:
Main objective: To evaluate the bidirectional relationships between physical exercise and sleep parameters, as a part of multimodal prehabilitation intervention, on pre- and postoperative outcomes in surgical patients with colorectal cancer, in an RCT.

Secondary objective: to determine whether the levels of anxiety and depression affect these relationships.

Objectives are based on the overarching hypothesis that is sleep and physical activity influence each other through complex, reciprocal interactions including multiple physiological and psychological pathways. To achieve this, providing a multimodal prehabilitation, specifically physical exercise, involved in mental and physical health through different mechanisms, i.e., improving physical functioning and fitness, reducing side effects of cancer treatments, preventing bone loss and weight gain, improving the quality of life and sleep, decreasing symptoms of fatigue and depression.

The present is a pilot study aiming to evaluate the bidirectional relationships between sleep and physical exercise, and the preliminary outcome has important implications for informing both clinical and public health practice.

Research question: Does a multimodal intervention including physical exercise improve sleep quality and duration compared to standard of care, during the perioperative period? Conversely, does a better sleep quality and duration increases the level of physical exercise during the perioperative period? How the level of anxiety and depression will affect these relationships? If the Prehabilitation program specifically physical exercise will positively affect sleep quality and duration after surgery, in the way to be a protective factor of sleep to not be reduced by up to 55% compared to those receiving standard of care?

DETAILED DESCRIPTION:
Participants will be referred by colorectal surgery of the MUHC-Montreal General Hospital; 100 participants will be studied. Inclusion: adult patients aged 18 years and older, of either sex undergoing colorectal cancer surgery. All adult persons scheduled for resection of malignant colorectal lesions will be included. Exclusion criteria: a compromised health status (American Society of Anesthesiologists [ASA] class 4-5) or comorbid medical conditions interfering with the ability to perform an exercise. Patients are unable to understand the information given, insufficient understanding of English or French language to provide informed consent or who are considered unable to perform study-specific procedures. Patients that diagnosis of a sleep disorder other than insomnia (e.g., sleep-disordered breathing) or received psychotherapy specifically for insomnia, as well as a night-shift worker in the past 3 months or the next 18 months will be excluded.

Study Design: Randomized controlled trial of two parallel arms: prehabilitation program and standard of care (SOC). Informed consent forms will be signed and dated before the conduct of any study-specific procedures. After baseline assessment, participants will be random, by a computer program, allocated to either an intervention or a control group. Duration and follow-up. The intervention will last for 4 weeks pre- and 8 weeks post-surgery, for a total of 12 weeks. Site visits will occur weekly before surgery and every 4 weeks after surgery. In that period, weekly phone calls will reinforce compliance and provide tips to help patients adhere to the treatment protocol. A dedicated and specially trained research team lead by a physician, a kinesiologist, a nutritionist and a psychologist will perform the measurements and collect the demographic and surgical details of all the patients, recording daily detailed information of clinical outcomes up to 8 weeks after surgery.

Interventions: Common to both groups: as part of the enhanced recovery after surgery (ERAS) protocol as the standard of care in our institution. All participants will wear an actigraphy to objectively assess their daily physical activity and their sleep behavior. The following outcomes will be assessed for all participants, at the baseline and will be repeated after 4 weeks, before and after the surgery: sleep behaviors included sleep quality and duration, assessed subjectively and objectively. Self-reported and objective outcome measurements will be assessed from all participants such as the 6-minute walk distance (6MWD), daily activity counts, exercise tolerance (CPET) and handgrip strength, Insomnia Severity Index (ISI), Chronotype, health-related quality of life assessed by using the Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36) and the Hospital Anxiety and Depression Scale (HADS) used to assess emotional distress.

ELIGIBILITY:
Inclusion Criteria:

* All adult persons scheduled for resection of malignant colorectal lesions will be included

Exclusion Criteria:

* A compromised health status (American Society of Anesthesiologists [ASA] class 4-5) or comorbid medical conditions interfering with the ability to perform an exercise.
* Patients are unable to understand the information given, insufficient understanding of English or French language to provide informed consent or who are considered unable to perform study-specific procedures.
* Patients that diagnosis of a sleep disorder other than insomnia (e.g., sleep-disordered breathing) or received psychotherapy specifically for insomnia, as well as a night-shift worker in the past 3 months or the next 18 months will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-09-15 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI): "change" is being assessed | At the baseline, it will be repeated the week of the surgery and at 4 and 8 weeks after the surgery.
  This questionnaire was developed to assess the global subjective sleep disturbances of the previous month. The PSQI is a 19-item self-report measure of broad sleep disturbances over the past month and yields 7 component scores (subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, and daytime dysfunction), which are added to create a total score. Each score ranging from 0 to 3 and a total score range of 0-21, a score of 0 indicated no sleep problems and 3 indicated serious sleep problems.
Sleep quality by an Actigraphy: "change" is being assessed | 4 weeks before surgery and 4 weeks after the surgery
  Sleep quality will be objectively measured using the Actiwatch-2. The Actiwatch-2 (Philips, Respironics) is a small, waterproof, non-intrusive actigraphy device that is worn on the wrist of the non-dominant hand. By calculating orientation and movement, actigraphy records sleep-wake activity and provide an objective measure of sleep quality.

SECONDARY OUTCOMES:
Community Health Activities Model Program for Seniors (CHAMPS) questionnaire: "change" is being assessed | At the baseline, it will be repeated the week of the surgery and at 4 and 8 weeks after the surgery.
  The CHAMPS is a self-reported measure of physical activity, comprising 41 activities evaluated according to the total number of hours done during an average week. The CHAMPS has been validated as a measure of increasing levels of physical activity in older adults.
  1 METs), low-light (ie, > 1 and ≤2 METs; eg, playing cards), high-light (ie, >2 and <3 METs; eg, light walking), moderate-to-vigorous physical activity (MVPA, ≥3 METs), and "total activity" (≥2 METs)
Daily activity counts measured by an Actigraphy: "change" is being assessed | 4 weeks before surgery and 4 weeks after the surgery
  The Actiwatch-2 (Philips, Respironics) provide an objective measure of the daily activity counts.
Functional capacity using the six-minute walk test (6MWT): "change" is being assessed | At the baseline, it will be repeated the week of the surgery and at 4 and 8 weeks after the surgery.
  The 6MWT evaluates the ability to maintain a moderate level of physical activity reflecting the activities of daily living. Norms available: The six-minute walk distance in healthy adults has been reported to range from 400m to 700m. A lower score (reflecting less distance covered in 6 minutes) indicates worse function.
Hospital Anxiety and Depression Scale (HADS): "change" is being assessed | At the baseline, it will be repeated the week of the surgery and at 4 and 8 weeks after the surgery.
  The HADS contains seven items, each scored from 0 to 3 points for anxiety and depression. It provides summary measures on a scale of 0-21, with scores exceeding 8 suggesting the presence of a mood disorder.

OTHER OUTCOMES:
Insomnia Severity Index (ISI): "change" is being assessed | At the baseline, it will be repeated the week of the surgery and at 4 and 8 weeks after the surgery.
  To report the perceived severity of difficulties falling asleep, difficulties maintaining sleep and early morning awakenings, as well as the degree of dissatisfaction with current sleep, the degree to which sleep difficulties interfere with daytime functioning, the degree to which the deterioration of functioning related to the sleep problem is noticeable by others, and the level of distress or worry caused by the sleep difficulties.
  The total score is interpreted as follows: the absence of insomnia (0-7); sub-threshold insomnia (8-14); moderate insomnia (15-21); and severe insomnia (22-28).
Chronotype: "change" is being assessed | At the baseline, it will be repeated the week of the surgery and at 4 and 8 weeks after the surgery.
  One hears about 'morning' and 'evening' types of people with 5 response categories.
Health-related quality of life will be assessed using the Medical Outcomes Study 36-Item: "change" is being assessed Short-Form Health Survey (SF-36) | At the baseline, it will be repeated the week of the surgery and at 4 and 8 weeks after the surgery.
  A reliable and valid generic index of perceived health status for cancer patients and used on the previous study for patients undergoing scheduled colorectal surgery. 36-item patient-reported questionnaire that covers eight health domains: physical functioning (10 items), bodily pain (2 items), role limitations due to physical health problems (4 items), role limitations due to personal or emotional problems (4 items), emotional well-being (5 items), social functioning (2 items), energy/fatigue (4 items), and general health perceptions (5 items). Scores for each domain range from 0 to 100, with a higher score defining a more favorable health state.
The World Health Organization Disability Assessment Schedule (WHODAS 2.0): "change" is being assessed | At the baseline, it will be repeated the week of the surgery and at 4 and 8 weeks after the surgery.
  12 items used to measures disability due to health conditions including diseases, illnesses, injuries, mental or emotional problems, and problems with alcohol or drugs.
  The sum score for global disability therefore ranges from 0 (no disability) to 48 (complete disability).
Patient-Generated Subjective Global Assessment (PG-SGA): "change" is being assessed | At the baseline, it will be repeated the week of the surgery and at 4 and 8 weeks after the surgery.
  Validated for oncologic patients, it comprises 4 scored domains: recent weight loss, food intake, symptoms, and activities and functions. PG-SGA Short Form is a patient-reported instrument for the assessment of nutrition status in patients with cancer. The PG-SGA Short Form numerical scoring range from 0 (no problems) to 36 (worst problem).
The oxygen peak during cardiopulmonary exercise testing (CPET): "change" is being assessed | At the baseline, it will be repeated the week of the surgery and at 4 and 8 weeks after the surgery.
  CPET has a growing role in major abdominal surgery to guide decision-making by clinicians and to evaluate the consequences of neo-adjuvant therapies and prehabilitation programs.
  The term 'peak VO2' is used as a synonym for VO2 max throughout this text. Peak VO2 is considered abnormal when below 85% of the predicted value.
Anaerobic threshold (AT) measured during cardiopulmonary exercise testing (CPET): "change" is being assessed | At the baseline, it will be repeated the week of the surgery and at 4 and 8 weeks after the surgery.
  The VO2 value measured in the first ventilatory threshold (VT1) or anaerobic threshold (AT) is determined by the nonlinear increase of pulmonary ventilation (VE) in relation to VO2. The normal mean AT values expected for adults is around 40% to 65% of peak VO2.
Pulmonary ventilation measured during cardiopulmonary exercise testing (CPET): "change" is being assessed | At the baseline, it will be repeated the week of the surgery and at 4 and 8 weeks after the surgery.
  Pulmonary ventilation (VE): Ventilation increases continuously during progressive effort on CPET and undergoes additional increases influenced by the anaerobic metabolism resulting from the accumulation of lactic acid, well defined as the first and second ventilatory thresholds. Periodic (or oscillatory) ventilation is defined as the resting oscillatory pattern that persists in ≥ 60% of the effort with an amplitude of ≥ 15% as compared to mean resting values.
CO2 production: "change" is being assessed | At the baseline, it will be repeated the week of the surgery and at 4 and 8 weeks after the surgery.
  CO2 production measured during cardiopulmonary exercise testing (CPET)
O2 consumption: "change" is being assessed | At the baseline, it will be repeated the week of the surgery and at 4 and 8 weeks after the surgery.
  O2 consumption measured during cardiopulmonary exercise testing (CPET)
Respiratory coefficient measured during cardiopulmonary exercise testing (CPET): "change" is being assessed | At the baseline, it will be repeated the week of the surgery and at 4 and 8 weeks after the surgery.
  Respiratory coefficient or respiratory exchange ratio (R): expresses the ratio between CO2 production and O2 consumption (VCO2/VO2). It is currently the best non-invasive indicator of maximal or quasi-maximal exercise intensity. Values above 1.0 can reflect intense exercise, but those ≥ 1.10 are those searched on CPET, and have been accepted as a parameter of exhaustion or quasi-exhaustion.
Muscle strength Handgrip strength will be measured with the Jamar hydraulicdynamometer, in kg: "change" is being assessed | At the baseline, it will be repeated the week of the surgery and at 4 and 8 weeks after the surgery.
  Maximal strength will be recorded, according to standardized procedures. Isokinetic leg strength will be measured with a Biodex on the dominant side.
  Loss of muscle strength was defined as < 30kg (men) and < 20 kg (women).
Height: "change" is being assessed | At the baseline, it will be repeated the week of the surgery and at 4 and 8 weeks after the surgery.
  Height with a ruler on the wall measured in cm
Weight: "change" is being assessed | At the baseline, it will be repeated the week of the surgery and at 4 and 8 weeks after the surgery.
  Bodyweight will be measured by a digital scale by the Seca mBCA machine in kg

CONTACTS AND LOCATIONS:
Overall Officials: Sender Liberman, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Franco Carli, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Davies NJ, Batehup L, Thomas R. The role of diet and physical activity in breast, colorectal, and prostate cancer survivorship: a review of the literature. Br J Cancer. 2011 Nov 8;105 Suppl 1(Suppl 1):S52-73. doi: 10.1038/bjc.2011.423. PMID 22048034
- [Background] Meyerhardt JA, Giovannucci EL, Holmes MD, Chan AT, Chan JA, Colditz GA, Fuchs CS. Physical activity and survival after colorectal cancer diagnosis. J Clin Oncol. 2006 Aug 1;24(22):3527-34. doi: 10.1200/JCO.2006.06.0855. Epub 2006 Jul 5. PMID 16822844
- [Background] Albrecht TA, Taylor AG. Physical activity in patients with advanced-stage cancer: a systematic review of the literature. Clin J Oncol Nurs. 2012 Jun 1;16(3):293-300. doi: 10.1188/12.CJON.293-300. PMID 22641322
- [Background] Carli F, Charlebois P, Stein B, Feldman L, Zavorsky G, Kim DJ, Scott S, Mayo NE. Randomized clinical trial of prehabilitation in colorectal surgery. Br J Surg. 2010 Aug;97(8):1187-97. doi: 10.1002/bjs.7102. PMID 20602503
- [Background] Mayo NE, Feldman L, Scott S, Zavorsky G, Kim DJ, Charlebois P, Stein B, Carli F. Impact of preoperative change in physical function on postoperative recovery: argument supporting prehabilitation for colorectal surgery. Surgery. 2011 Sep;150(3):505-14. doi: 10.1016/j.surg.2011.07.045. PMID 21878237
- [Result] Chen HM, Tsai CM, Wu YC, Lin KC, Lin CC. Effect of walking on circadian rhythms and sleep quality of patients with lung cancer: a randomised controlled trial. Br J Cancer. 2016 Nov 22;115(11):1304-1312. doi: 10.1038/bjc.2016.356. Epub 2016 Nov 3. PMID 27811855
- [Result] Romain B, Rohmer O, Schimchowitsch S, Hubner M, Delhorme JB, Brigand C, Rohr S, Guenot D. Influence of preoperative life satisfaction on recovery and outcomes after colorectal cancer surgery - a prospective pilot study. Health Qual Life Outcomes. 2018 Jan 17;16(1):16. doi: 10.1186/s12955-017-0824-4. PMID 29343246
- [Result] Lin KY, Shun SC, Lai YH, Liang JT, Tsauo JY. Comparison of the effects of a supervised exercise program and usual care in patients with colorectal cancer undergoing chemotherapy. Cancer Nurs. 2014 Mar-Apr;37(2):E21-9. doi: 10.1097/NCC.0b013e3182791097. PMID 23357886
- [Result] Coles T, Bennett AV, Tan X, Battaglini CL, Sanoff HK, Basch E, Jensen RE, Reeve BB. Relationship between sleep and exercise as colorectal cancer survivors transition off treatment. Support Care Cancer. 2018 Aug;26(8):2663-2673. doi: 10.1007/s00520-018-4110-8. Epub 2018 Feb 22. PMID 29470704
- [Result] Cho MH, Dodd MJ, Cooper BA, Miaskowski C. Comparisons of exercise dose and symptom severity between exercisers and nonexercisers in women during and after cancer treatment. J Pain Symptom Manage. 2012 May;43(5):842-54. doi: 10.1016/j.jpainsymman.2011.05.016. Epub 2012 Mar 19. PMID 22436836
- [Result] Brunet J, Burke S, Grocott MP, West MA, Jack S. The effects of exercise on pain, fatigue, insomnia, and health perceptions in patients with operable advanced stage rectal cancer prior to surgery: a pilot trial. BMC Cancer. 2017 Feb 23;17(1):153. doi: 10.1186/s12885-017-3130-y. PMID 28228123
- [Result] Cheville AL, Kollasch J, Vandenberg J, Shen T, Grothey A, Gamble G, Basford JR. A home-based exercise program to improve function, fatigue, and sleep quality in patients with Stage IV lung and colorectal cancer: a randomized controlled trial. J Pain Symptom Manage. 2013 May;45(5):811-21. doi: 10.1016/j.jpainsymman.2012.05.006. Epub 2012 Sep 24. PMID 23017624
- [Result] Young-McCaughan S, Mays MZ, Arzola SM, Yoder LH, Dramiga SA, Leclerc KM, Caton JR, Sheffler RL, Nowlin MU. Research and commentary: Change in exercise tolerance, activity and sleep patterns, and quality of life in patients with cancer participating in a structured exercise program. Oncol Nurs Forum. 2003 May-Jun;30(3):441-54; discussion 441-54. doi: 10.1188/03.ONF.441-454. PMID 12719744
- [Result] Rabin C, Pinto B, Dunsiger S, Nash J, Trask P. Exercise and relaxation intervention for breast cancer survivors: feasibility, acceptability and effects. Psychooncology. 2009 Mar;18(3):258-66. doi: 10.1002/pon.1341. PMID 18473397